CLINICAL TRIAL: NCT03774966
Title: Do Patients Who Receive the IPACK and Adductor Canal Catheter Have Better Outcomes Than Patients Receiving the Adductor Canal Catheter Alone for Total Knee Replacements?
Brief Title: IPACK and Adductor Canal Catheter Patient Outcomes for TKAs?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Eva Boyd, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-001490
Record Dates: First submitted 2018-12-04; First posted 2018-12-13 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Surgery; Acute Pain
Keywords: total knee arthroplasty; regional block
MeSH Terms: conditions — Acute Pain | interventions — Catheters

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adductor Canal Block + Catheter (Active Comparator): Adductor canal block: 15 mL of 0.25% ropivicaine, adductor canal catheter: 6 mL/hr of 0.2% ropivacaine
  Interventions: Procedure: Adductor canal block + catheter
- Adductor Canal Block + Catheter & IPACK (Experimental): Adductor canal block: 15 mL of 0.25% ropivicaine, adductor canal catheter: 6 mL/hr of 0.2% ropivacaine, IPACK block: 15 ml of 0.25% ropivacaine.
  Interventions: Procedure: Adductor Canal Block + Catheter & IPACK block

INTERVENTIONS:
Procedure: Adductor Canal Block + Catheter & IPACK block — Adductor Canal Block + Catheter & IPACK block
  Arms: Adductor Canal Block + Catheter & IPACK
Procedure: Adductor canal block + catheter — Adductor canal block + catheter
  Arms: Adductor Canal Block + Catheter

SUMMARY:
This study evaluates the addition of the IPACK block to the adductor canal block and catheter in the pain management of total knee arthroplasty. Half of participants will receive the adductor canal block and catheter with the IPACK block, while the other half will receive the adductor canal block and catheter only.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a surgical procedure that can be associated with significant post-operative pain. Poor pain control in the post-operative period has contributed to delays in early mobility and rehabilitation, an important part of recovery that is best started as soon as possible after surgery. Regional techniques in general have helped manage post-operative pain as well as minimize narcotic use. The application of femoral and sciatic nerve blocks has been shown to decrease opioid use; however, they were associated with adverse events such as quadriceps weakness and falls post-operatively. This led to the development of the adductor canal block (ACB) which has gained favor for providing superior analgesia over opioids alone, and for the added benefit of sparing the quadriceps muscle. Recently, adding local anesthetic to the interspace between the popliteal artery and posterior capsule of the knee (IPACK) blocks have been used to help address pain in the posterior part of the knee that is not well covered by the adductor canal block alone. While the sciatic nerve block is also an option to cover this area, it is associated with foot drop which can hinder early mobility. For patients undergoing TKAs at UCLA, our standard of practice is the ACB. The investigators hope to show with this study that adopting this novel block will help with post-operative pain control, decrease length of hospital stay, and increase distance walked during physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee replacement without contraindications to regional blocks

Exclusion Criteria:

* Patients who have contraindications to regional blocks: infection at injection site for the nerve block, allergy to local anesthetics, history of a bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in milligram morphine equivalents | 4 days
  Total opioid consumption will be calculated for postoperative day 0-3 ( postoperative day 0 is the day of the surgery and is the first day of the time frame and postoperative day 3 is the 4th day) and total hospital stay. Opioid amount will be converted to morphine equivalents (milligram) for comparison.

SECONDARY OUTCOMES:
Visual analog pain scores | 4 days
  Pain scores will be assessed postoperative day 0-3 ( postoperative day 0 is the day of the surgery and is the first day of the time frame and postoperative day 3 is the 4th day) using the visual analog score (Scale 0-10). Zero for no pain and ten being the worst pain experienced. They will be obtained and recorded every 4 to 6 hours by the nurse monitoring the subject.
Distance ambulated during physical therapy | 4 days
  Distance (meters) ambulated during physical therapy will be recorded for postoperative day 0-3 ( postoperative day 0 is the day of the surgery and is the first day of the time frame and postoperative day 3 is the 4th day)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Medical Center, Santa Monica, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cullom C, Weed JT. Anesthetic and Analgesic Management for Outpatient Knee Arthroplasty. Curr Pain Headache Rep. 2017 May;21(5):23. doi: 10.1007/s11916-017-0623-y. PMID 28283810
- [Result] Thobhani S, Scalercio L, Elliott CE, Nossaman BD, Thomas LC, Yuratich D, Bland K, Osteen K, Patterson ME. Novel Regional Techniques for Total Knee Arthroplasty Promote Reduced Hospital Length of Stay: An Analysis of 106 Patients. Ochsner J. 2017 Fall;17(3):233-238. PMID 29026354